CLINICAL TRIAL: NCT02283437
Title: A Randomized Controlled Trial of Problem-solving Based Bibliotherapy Program for Family Caregivers of People With Schizophrenia Spectrum Disorders
Brief Title: A Problem-solving Based Bibliotherapy Program for Family Caregivers in Schizophrenia
Acronym: PSBPF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Integrated Community Care and Family Support Centres (Unknown)
Responsible Party: Principal Investigator, Prof. Wai Tong CHIEN, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HSEARS2014218003
Record Dates: First submitted 2014-11-03; First posted 2014-11-05 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Schizophrenia Spectrum Disorders; Family Caregivers
Keywords: Bibliotherapy; Problem-solving; Randomized Controlled Trial; Schizophrenia Spectrum Disorders; Family Caregivers

STUDY DESIGN:
Intervention Model Description: Repeated-measures, three-arm design
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors are blind to the group assignment and intervention received by the participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Problem-solving Based Bibliotherapy (Experimental): The Problem-solving Based Bibliotherapy Program (PSBPF) using a self-help manual based on problem-solving therapy defined by D'Zurilla and Nezu (2007) to be 'a self-directed cognitive-behavioral process by which a person attempts to identify/discover effective/adaptive solutions for specific problems encountered in everyday living' (p.11).
  Interventions: Behavioral: Problem-solving Based Bibliotherapy Program
- Behavioral Management and Education Program (Active Comparator): The Behavioral Management and Education group program will be guided by a validated treatment protocol based on the research team's (Chien and Wong, 2007) psycho-education and McFarlane et al.'s (2003) family behavioral management programs for schizophrenia.
  Interventions: Behavioral: Behavioral Management and Education Program
- Routine Outpatient Service (No Intervention): Participants in the control group (and 2 treatment groups) will receive routine psychiatric outpatient and family services.

INTERVENTIONS:
Behavioral: Problem-solving Based Bibliotherapy Program — The PSBPF will complete the bibliotherapy (self-help) and problem-solving manual developed by the research team for caregivers of people with schizophrenia spectrum disorders.
  Other Names: PSBPF
  Arms: Problem-solving Based Bibliotherapy
Behavioral: Behavioral Management and Education Program — Two trained advanced practice psychiatric nurses who are experienced in psychiatric rehabilitation and group programs will lead the behavioral management and education group, which is guided by a validated treatment protocol based on the research team's (Chien and Wong, 2007) and McFarlane et al.'s (2001) family management programs for schizophrenia.
  Arms: Behavioral Management and Education Program

SUMMARY:
This proposed randomized controlled trial will test the effectiveness of a problem-solving based bibliotherapy program (PSBPF) for Chinese family caregivers in schizophrenia spectrum disorders. A repeated-measures, three-group design will be used to evaluate and compare the effects between two treatment groups (PSBPF and behavioral management group) and routine outpatient service (control group) for 150 randomly selected family caregivers of outpatients with schizophrenia-spectrum disorders over a 18-month follow-up.

DETAILED DESCRIPTION:
Family caregivers of people with schizophrenia-spectrum disorders are confronted by a various physical, psychosocial and financial hardships. This can adversely affect family members' caregiving experiences, psychological distress, general well-being, and family relationships or emotional involvement, which in turn may contribute to a greater risk of patient relapse and non-recovery. While family psycho-education (behavioral management) and mutual support groups are effective in reducing caregivers' burden of care, these approaches usually require regular meetings and encounter difficulties in extensive training of group leaders/facilitators and engaging participants to actively share their caregiving experiences due to time inconvenience and fear/inability of expression of feelings. By virtue of the above, an alternate model of self-help program in book form named bibliotherapy, which is a guided reading and self-practice program with problem-solving training facilitated by a psychiatric nurse, has recently demonstrated evidences in clinical trials for families of depressive and psychotic patients by the research team, and other researchers.

This proposed randomized controlled trial will test the effectiveness of a problem-solving based bibliotherapy program (PSBPF) for Chinese family caregivers in schizophrenia spectrum disorders. A repeated-measures, three-group design will be used to evaluate and compare the effects between two treatment groups (PSBPF and behavioral management and educational group) and routine outpatient service and family support(control group) for 150 randomly selected family caregivers of outpatients with schizophrenia-spectrum disorders over a 18-month follow-up. Primary outcomes include caregivers' burden of care, caregiving experiences and coping and social problem-solving skills using validated instruments. Secondary outcomes are patients' mental state, functioning, perceived expressed emotion, and re-hospitalization rate. They will be measured at recruitment, one week, and 6 and 18 months following the interventions. Kaplan-Meier survival analysis will be used to analyze the relative risks of re-hospitalizations amongst the treatment and control groups over 18-month follow-up. It is hypothesized that the PSBPF participants will produce significantly better improvements in caregivers' perceived burden, caregiving experience and coping and problem-solving skills than those in behavioral management/education and control groups over 18-month follow-up.

Focus group interviews will be conducted after the first post-test with 30 caregivers (15 participants per group) in both treatment groups. Their data will be content analyzed to identify their perceived benefits, limitations and difficulties encountered and therapeutic ingredients of the two programs. With significant positive outcomes found in the PSBPF, this program will be adopted by community mental healthcare services in Hong Kong, and replicated in other Asian countries, to improve family-based care in schizophrenia-spectrum disorders.

Study Objectives:

This controlled trial tests the effects of the PSBPF on family caregivers' and patients' outcomes over a 18-month follow-up, when compared with those in a behavioral management and education group or routine family services for outpatients. Primary outcomes include caregivers' burden of care, coping and problem-solving skills. It will test two hypotheses that, comparing with those in behavioral management and education/routine care, the PSBPF will indicate significantly:

* greater reduction of caregivers' perceived burden and improvements in coping and social problem-solving skills and caregiving experiences at 1-week, 6-month and/or 18-month follow-ups; and
* greater improvements in patients' mental state, psychosocial functioning, perceived expressed emotion, and re-hospitalization rate at the three follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong Chinese residents, aged 18-64;
* Taking care of a family member primarily diagnosed as schizophrenia spectrum disorders, including schizophrenia, schizophreniform and schizoaffective disorders, as stated in the criteria of the Diagnostic and Statistical Manual (DSM-IV Text-Revised edition) in the past 3 years;
* Able to read and understand Cantonese/Mandarin; and
* Perceived a moderate to high burden of care (measured by Family Burden Interview Schedule (>20 out of 50 scores for case selection).

Exclusion Criteria:

* Caregivers have received or are receiving another family intervention; or
* Presented with a recent personal history of a serious mental illness/medical disease and/or learning difficulties.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Perceived Burden of Care | 18 months after completion of intervention
  Caregivers' perceived burden of care will be measured by a Chinese version of the 25-item Family Burden Interview Schedule. It assesses the caring burden perceived by family members in taking care of the patient at home. It is comprised of six categories (2-6 items per category), including familial finance, routine, leisure activities, interactions, and physical and mental health. Total scores range from 0-50; a higher score will indicate a greater caring burden. The Chinese version of the scale indicated satisfactory internal consistency (Cronbach's alpha= 0.87) and high inter-rater reliability (Pearson's r= 0.75-0.99) in families of schizophrenia sufferers in Hong Kong.
Coping Style | 18 months follow-up
  A Chinese version of Coping style of the caregivers style will be assessed using the 42-item Revised Ways of Coping Checklist. It composes of a problem-focused coping(15 items) and three emotion-focused coping scales, including 'self-blame' (3 items), 'wishful thinking'(8 items) and 'avoidance'(10 items), and a subscale 'seeking social support'(6 items). Items are scored on a 5-point Likert scale, from '0-never' to '4-all the time', higher scores indicating greater uses of those coping strategies. It has demonstrated satisfactory internal consistency (Cronbach's alpha= 0.62-0.85) in students.
Social Problem-Solving Inventory | 18 months follow-up
  The Chinese version of Revised (Short) Social Problem-Solving Inventory. It contains 25 items, assessing 2 domains of social problem-solving, including problem-solving style(3 subscales- rational problem solving, impulsive/careless style and avoidance style), and problem-solving orientation (2 subscales- positive and negative problem orientation). It has demonstrated satisfactory internal consistency (Cronbach's alpha= 0.68-0.81) and concurrent validity with a few coping scales in Hong Kong adolescents.[

SECONDARY OUTCOMES:
Experience of Caregiving | 18 months follow-up
  The Chinese version of Experience of Caregiving Inventory is a 66-item self-reporting scale that measures experiences of caregiving to a family member with mental illness based on the Transactional model of stress-appraisal-coping. It consists of 10 subscales measuring negative (e.g., difficult behaviors, stigma and problems with services) and positive aspects (positive personal experience and aspects of relationship) of caregiving, being rated on a 5-point Likert scale ('0-never' to '4-nearly always'). It indicates satisfactory content validity and internal consistency (Cronbach's alpha= 0.60-0.85); higher scores on negative/positive (reverse-coded) subscale indicate a more negative appraisals.
Mental State | 18 months follow-up
  Patients' mental state will be evaluated by the Positive and Negative Syndrome Scale, a 30-item inventory assessing the absence/severity of psychotic symptoms across positive symptoms, negative symptoms and general psycho-pathology symptoms. Each item is scored on a scale, ranging from '1- absent' to '7- extreme', and the scale has demonstrated good inter-rater reliability (Intra-class correlation= 0.88) and good internal consistency (Cronbach's alpha= 0.87-0.93), and concurrent and predictive validity.
Patient Functioning | 18 months follow-up
  The 43-item Specific Level of Functioning Scale will be used to assess 3 functional domains for patients with schizophrenia, including physical functioning/personal care (12 items), social functioning (14 items) and community living skills (17 items) on a 5-point Likert scale. The Chinese version was validated among patients with schizophrenia in Hong Kong, indicating satisfactory content validity, test-retest reliability (Pearson's r=0.76) and internal consistency (Cronbach's alpha= 0.88-0.96).
Perceived Expressed Emotion | 18 months follow-up
  Perceived expressed emotion by patients will be measured by Level of Expressed Emotion scale. The scale comprises 4 domains: intrusiveness, attitude toward illness, tolerance/expectancy, and emotional responses; each consists of 15 items on a 4-point Likert scale ('1-Not true' to '4-True'). The Chinese version has indicated satisfactory internal consistency (Cronbach's alpha= 0.80-0.90) and test-retest reliability (r= 0.87-0.93)
Rate & Length of Rehospitalizations | 18 months follow-up
  The data of patients' frequency and lengths (days) of psychiatric hospitalizations over the intervention period, and 12-month follow-ups, will be recorded by the research assistant by reviewing the electronic patient record (ePR) at outpatient clinics.

CONTACTS AND LOCATIONS:
Overall Officials: Wai Tong Chien, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (2):
- Hong Kong (2):
  - KH OPD, Mong Kok, Kowloon
  - Li Ka Shing Specialty OPD, Shatin, NT

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McCann TV, Lubman DI, Clark E. First-time primary caregivers' experience of caring for young adults with first-episode psychosis. Schizophr Bull. 2011 Mar;37(2):381-8. doi: 10.1093/schbul/sbp085. Epub 2009 Aug 13. PMID 19679716
- [Background] McCann TV, Lubman DI, Cotton SM, Murphy B, Crisp K, Catania L, Marck C, Gleeson JF. A randomized controlled trial of bibliotherapy for carers of young people with first-episode psychosis. Schizophr Bull. 2013 Nov;39(6):1307-17. doi: 10.1093/schbul/sbs121. Epub 2012 Nov 20. PMID 23172001